CLINICAL TRIAL: NCT04065880
Title: Neoveil® Versus TachoSil® for the Treatment of Pulmonary Air Leaks Following Lung Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-01505; ch19Lardinois
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Prolonged Air Leak; Postoperative Air Leak
Keywords: lung resection; TachoSil®; Neoveil®; air leak closure; drainage time
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinded participants and unblinded investigators and evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TachoSil® (Active Comparator): TachoSil® is a collagen sponge coated with the human coagulation factors fibrinogen and thrombin.
  Interventions: Other: TachoSil®
- Neoveil® (Active Comparator): Neoveil® sheet made of polyglycolic acid (PGA). It is a biodegradable, thermoplastic and non-antigenic polymer.
  Interventions: Other: Neoveil®

INTERVENTIONS:
Other: TachoSil® — topical absorbable fibrin sealant patch applied directly on the lung area with air fistula.
  Arms: TachoSil®
Other: Neoveil® — bioabsorbable soft-tissue reinforcement material applied on the normal shape of the lung at the end of the operation.
  Arms: Neoveil®

SUMMARY:
Postoperative prolonged air leak (PAL), referring to the passage of air from the lung parenchyma into the pleural space, is one of the most frequent postoperative complications after lung resection. To control air leak, there are two different products certified since years: TachoSil® and Neoveil®. This study is to investigate the difference of TachoSil® and Neoveil® in patients with PAL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pulmonary air leak following open lung surgery, regardless of whether an anatomical or atypical resection was performed
* Patients who are able to decide for themselves whether to participate in the study or not ( for example due to language problems, mental disorders, dementia of the participant)
* Patients who are not family member or employee of the investigator

Exclusion Criteria:

* Inability to follow the procedures of the study, for example, due to language problems, mental disorders, dementia of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
time required till air leak closure has occurred (hours) | end of the operation (0 hours) until removal of the chest tubes or re-operation in case of prolonged air leak (first postoperative day)
  time interval between end of the operation (closure of the skin) and air leak closure (less than 30ml on the digitalized drainage system).

SECONDARY OUTCOMES:
Incidence of air leak (binary outcome 0/1), i.e. air loss > 30ml | end of the operation (0 hours) until removal of the chest tubes or re-operation in case of prolonged air leak (first postoperative day)
  Incidence of air leak (binary outcome 0/1), i.e. air loss > 30ml
Intensity of air leak (continuous outcome, ml) | end of the operation (0 hours) until removal of the chest tubes or re-operation in case of prolonged air leak (first postoperative day)
  Intensity of air leak (continuous outcome, ml)
Incidence of prolonged air leak (>10 days) (binary outcome 0/1) | assessed at 10th postoperative day
  Incidence of prolonged air leak (>10 days) (binary outcome 0/1)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. MD, Principal Investigator — Department of Thoracic Surgery, University Hospital Basel
Locations (1):
- Department of Thoracic Surgery, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Bachmann H, Dackam SVC, Hojski A, Jankovic J, Vogt DR, Wiese MN, Lardinois D. Neoveil versus TachoSil in the treatment of pulmonary air leak following open lung surgery: a prospective randomized trial. Eur J Cardiothorac Surg. 2022 Dec 2;63(1):ezad003. doi: 10.1093/ejcts/ezad003. PMID 36651370